CLINICAL TRIAL: NCT03382223
Title: Panel Study Investigating Status of Cognitively Impaired Elderly in Singapore
Acronym: PISCES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Chetna Malhotra, Assistant Professor, Duke-NUS Graduate Medical School
Other Study IDs: 2017/2989
Record Dates: First submitted 2017-12-07; First posted 2017-12-22 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Advanced Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dementia affects 10% of the elderly population in Singapore. However, there is a lack of systematic information regarding end of life (EOL) care received by patients dying with severe dementia (PDSD), PDSD's EOL direct and indirect costs and caregiver burden. This study, a first of-its-kind prospective cohort study in Singapore will assess the EOL care received by PDSD and PDSD's caregivers, EOL medical and social care costs of severe dementia and caregiver burden; and will develop a risk score to predict 6-month mortality for PDSD. The investigators will accomplish this by surveying caregivers of PDSD every 4 months till the patient passes away and 6 weeks and 6 months after patient's death during caregiver bereavement. The investigators will also extract and match patient medical and billing data with survey data for comprehensive assessment of care costs.

Key outcomes achieved by this study will be improved understanding of PDSD's EOL care, EOL care costs, and caregiver burden and bereavement. The systematic data collected will also lead to predicting 6 month mortality for community dwelling PDSD with greater accuracy compared to existing tools. Positive implications from this study will be improved early decision making by caregivers regarding EOL care and physician referrals for palliative care services; and a better understanding of EOL care for PDSD and PDSD's caregivers that will lead to cross-sector collaborations to improve delivery of palliative care to PDSD. In this way this proposal is highly responsive to the grant call which focuses on early decision making and cross sector palliative care delivery among non-cancer patients. In the long term, this study will improve clinical and public health policy and has the potential to be the foundation for future initiatives for dementia care and improved social and medical infrastructure planning.

ELIGIBILITY:
Inclusion Criteria for primary informal caregivers are:

1. Age ≥ 21 years old
2. Singaporean/Singapore Permanent Resident
3. Intact cognition determined through the Abbreviated Mental Test (AMT) for those who are ≥ 65 years old
4. Patients who score 20 or more on QDRS answered by caregivers will be considered to have severe dementia
5. Main person or one of the main persons providing care to patient (e.g. accompanying patient for doctor's visits, helping patient with day to day activities)
6. Main person or one of the main persons ensuring the provision of care to patient (e.g. supervision of foreign domestic worker so that patient is looked after)
7. Main person or one of the main persons involved in making decisions regarding treatment patient receives

Exclusion Criteria for primary informal caregivers are:

1. Caregivers ≥ 65 years old with cognitive impairment or serious mental illness determined through AMT
2. Foreign domestic workers/maids

Inclusion Criteria for physicians are:

(a) Caregivers of patients they are treating are enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study of primary informal caregivers of 400 patients dying with severe dementia (PDSD) who will be surveyed every 4 months for a period of 2 years or until the patient passes away and then post-death 6 weeks and 6 months to assess bereavement of the caregiver. Treating physicians of the patients will also be invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life of patient | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess the quality of life of patient by asking caregivers the list of comorbidities and acute medical conditions that patient has, patient's experience of symptoms, patient's functional status and behaviours that patient exhibits.
Change in quality of care received by patient | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess the quality of care received by patient by asking the caregiver of any use of tube-feeding, physical restraint and other medical interventions; as well as checking with the caregiver if they are satisfied with the care provided for patient.
Change in caregiver's resilience | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess caregiver's resilience through the abbreviated version of the Connor-Davidson Resilience Scale (CD-RISC), the CD-RISC 2. Only 2 items will be adapted from CD-RISC. For each item, it is rated on a 5-point scale, ranging from 0 to 4 as follows: "not true at all", "rarely true", "sometimes true", "often true" and "true nearly all of the time", with higher scores reflecting greater resilience.
Change in caregiver burden | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess caregiver burden through modified Caregiver Reaction Assessment (CRA) Instrument. This instrument captures 5 domains of caregiver reaction and we adopted 4 out of the 5 domains. Each item is scored on a five-point likert scale, ranging from 0 to 4 as follows: "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree". We amended and included "not applicable" to the scale as well. The items constituting a particular domain are averaged to generate subscale scores. A higher score on the subscales indicate greater negative effects of caregiving in those domains.
Change in caregiver's ability to cope | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess caregiver's ability to cope through the BriefCOPE instrument. This instrument measures 14 conceptually differentiable coping reactions; each of which comprises of 2 subscales. The scale ranges from 0 to 3 as follows: "I haven't been doing this at all", "I've been doing this a little bit", "I've been doing this a medium amount" and "I've been doing this a lot". This measure does not compute the overall score. The scales are analysed separately to see what its relation is to other variables.
Change in caregiver's levels of emotional distress | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess caregiver's anxiety and depression through the Hospital Anxiety and Depression Scale (HADS). The instrument comprises seven questions for anxiety and seven questions for depression. Each item comprises of a four point (0-3) response category. Hence the possible score ranges from 0 to 21 for anxiety and for depression. A score of 0 to 7 for either subscale is regarded as being in the normal range, a score of 11 or higher indicates probable presence of mood disorder and a score of 8 to 10 is suggestive of the presence of the respective state.
Change in caregiver's awareness of prognostic information | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess preferences of caregivers for the disclosure of prognostic information of patient.
Change in caregiver's grief experience | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess caregiver's grief experience through the MM Caregiver Grief Inventory- Short Form (MM-CGI-SF). The instrument consists of 3 domains (each domain has 6 items) with a total of 18 items. For each item, the scale ranges from 1 to 5 as follows: "strongly disagree", "disagree", "somewhat agree", "agree" and "strongly agree". The subscale is computed by summing up the scores of the 6 items for each domain. Higher scores may indicate a need for formal intervention or support assistance to enhance coping, while lower scores may indicate denial or a downplaying of distress or positive adaptation if the individual is not showing other signs of suppressed grief. The total grief level is computed by summing up the scores for the 18 items.The higher the score, the greater the level of grief experienced by the caregiver, vice versa.
Change in resource utilisation for patient | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will assess the healthcare resource utilisation of patient and caregiver through modified Resource Utilisation in Dementia Lite (RUD-Lite) Instrument.
Total healthcare expenditure during the last year of life through analysis of medical bills | From recruitment to death of patient (baseline, 4 month, 8 month, 12 month, 16 month, 20 month, 24 month)
  We will calculate total healthcare expenditure during the last year of patient's life as the sum total of expenditures incurred at in-patient clinics, out-patient clinics, and visits to emergency department and on prescription drugs.

SECONDARY OUTCOMES:
Caregiver's perception of patient's quality of life at end-of-life, assessed after patient's death | 6 weeks bereavement
  We will assess caregiver's perception of patient's end-of-life care after patient's death through the Satisfaction With Care at the End of Life in Dementia (SWC-EOLD) scale. The scale has 10 items, each measured on a 4-point likert scale ranging from 1 to 4 as follows: "strongly disagree", "disagree", "agree", "strongly agree". The total SWC-EOLD score is computed by the summation of all 10 items (range of 10 to 40), with higher scores indicating more satisfaction.
Caregiver's bereavement adjustment | 6 months bereavement
  Post-patient death bereavement adjustment will be assessed through the Brief Grief Questionnaire. This is a 5-item interview instrument for screening complicated grief. For each item, the scale ranges from 0 to 2 as follows: "not at all", "somewhat" and "a lot". The total score is computed by summing up the score for each item. If the total score is 5 or more, it may be suggestive of the presence of the syndrome of complicated grief.
Cultural stigma associated with dementia | Up to 6 months post-bereavement
  We will assess the cultural stigma associated with dementia by asking in-depth questions such as caregiver's perception of dementia before and after patient's diagnosis, caregiver's experience of outsiders' responses and attitudes towards dementia and how physicians give the diagnosis of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Chetna Malhotra, MD, MPH, Principal Investigator — Lien Centre for Palliative Care/Duke-NUS Medical School
Locations (9):
- Singapore (9):
  - Tsao Foundation, Singapore
  - Singapore General Hospital, Singapore
  - Alzheimer's Disease Association, Singapore
  - Care for the Elderly Foundation, Singapore
  - Changi General Hospital, Singapore
  - Institute of Mental Health, Singapore
  - Jurong Community Hospital, Singapore
  - St. Luke's Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore

REFERENCES:
- [Derived] Malhotra C, Chaudhry I, Shah SU, Ostbye T, Malhotra R. Trajectories of negative and positive experiences of caregiving for older adults with severe dementia: application of group-based multi-trajectory modelling. BMC Geriatr. 2024 Feb 19;24(1):172. doi: 10.1186/s12877-024-04777-w. PMID 38373922
- [Derived] Malhotra C, Vishwanath P, Yong JR, Ostbye T, Seow D, Yap P, Tan LL, Tham WY, Vaingankar J, Foo J, Tan BY, Tong K, Ng WC, Allen JC Jr, Malhotra R, Tan WM, Wee SL, Ng LL, Goveas R, Mok V, Sim A, Ng WF, Wong HK, Balasundaram B, Tan RQ, Ong PS, Cheong CY, Yee Chung Pheng A, Tiong C, Hum A, Lee A, Finkelstein EA. A Prospective Longitudinal Study of Caregivers of Community Dwelling Persons with Severe Dementia (PISCES): Study Protocol. J Alzheimers Dis. 2020;75(2):403-416. doi: 10.3233/JAD-190897. PMID 32280086